CLINICAL TRIAL: NCT03412604
Title: Effect of Modulating Gamma Oscillations by Transcranial Alternating Current Stimulation on Brain Structure and Function in Humans
Brief Title: Effect of Modulating Gamma Oscillations Using tACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Defense Advanced Research Projects Agency (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emiliano Santarnecchi, Associate Professor of Radiology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017P000648
Record Dates: First submitted 2018-01-22; First posted 2018-01-26 (Actual); Results first posted 2021-05-21 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- tACS (Experimental): Transcranial alternating current stimulation (tACS) tuned at the frequency of 40Hz (gamma frequency) will be applied for 1 hour in 20 sessions on consecutive weekdays. The tACS intervention (20 sessions) will be preceded and followed by amyloid, microglia and tau PET imaging as well as a clinical/cognitive evaluation. The assessment of the effect of stimulation on microglia activation, amyloid deposition and tau deposition will constitute a primary outcome measure. Assessment of adverse effects will be also evaluated as a secondary outcome. The effect of brain stimulation on brain connectivity will be assessed by EEG and MRI and cognitive function.
  Interventions: Device: Transcranial Alternating Current Stimulation (tACS)

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation (tACS) — tACS will be applied at a frequency of 40Hz and targeting the area of maximal tracer uptake on amyloid PET imaging using an individualized multielectrode design to maximize the induced electrical current to the target region.
  Other Names: Non-invasive Brain Stimulation

SUMMARY:
This study aims to implement an intervention based on multiple, individualized multifocal tACS stimulation sessions based on individual PET and MRI information in patients with amyloid-positive PET with the hope that this leads to microglia activation and decrease in cerebral amyloid and tau depositions in human patients with AD.

DETAILED DESCRIPTION:
This study will leverage all this accumulated knowledge by implementing an intervention based on multiple, individualized multifocal tACS stimulation sessions based on individual PET and MRI information in patients with amyloid-positive PET with the hope that this leads to microglia activation and decrease in cerebral amyloid and tau depositions in human patients with AD.This would have immense translational impact, as gamma tACS is an intervention that is portable, does not require expensive hardware, can be widely applied to large numbers of patients with AD, as well as, given its favorable side effect profile, even to patients at earlier stages of the disease who have cerebral amyloid/tau without clinical symptoms.

The investigators aim to enroll 10 individuals with AD with evidence of increased cerebral amyloid burden on amyloid PET imaging. This would allow for a final sample size of 5-6 fully evaluable subjects. Each subject's participation in this study will consist of approximately 31-35 visits: 1 day for consent and screening procedures, 5-7 days of baseline procedures (this includes the PET scans), 20 tACS study visits, and 5-7 days of follow-up assessments. Subjects will undergo baseline cognitive assessment, structural and functional MRI characterization, PET imaging to assess amyloid burden, tau deposition and level of microglia activation, and resting-state EEG measurement. Additionally, subjects will undergo a TMS-EEG and a tACS-EEG recording session to assess brain plasticity levels and identify markers of response to stimulation. All subjects will subsequently undergo 20 sessions of gamma-frequency (40 Hz) tACS. At the end of the 20 sessions, subjects will then repeat the baseline assessments over 5-7 visits, including repeat PET imaging to assess for changes in amyloid burden, tau deposition, and microglia activation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of mild to moderate AD*
* Mini Mental State Examination (MMSE) > 18
* Mild AD ≥ 21
* Moderate AD 18-20
* Demonstration or history of memory impairments.

  * Confirmation of diagnosis will be made by the study MD based on a holistic consideration of the participant's cognitive evaluation and history.
* Amyloid positive PET imaging
* At least 45 years old
* On a stable dose of medications for memory loss including cholinesterase inhibitors (e.g. donepezil, rivastigmine or memantine) as defined as 6 consecutive weeks of treatment at an unchanging dose
* Minimum of completed 8th grade education
* IQ> 85 as determined by the WTAR and no history of intellectual disability

Exclusion Criteria:

* Current history of poorly controlled migraines including chronic medication for migraine prevention
* Current or past history of any neurological disorder other than dementia, such as epilepsy, stroke, progressive neurologic disease (e.g. multiple sclerosis) or intracranial brain lesions; and history of previous neurosurgery or head trauma that resulted in residual neurologic impairment.
* Past or current history of major depression, bipolar disorder or psychotic disorders, or any other major psychiatric condition.
* Contraindication for undergoing MRI or receiving TMS or tACS,
* >50 mSv of radiation exposure for research within the past year (PET imaging exclusion)
* Presence of the Thr/Thr polymorphism in the TSPO gene (rs6971) due to low affinity binding for the PBR 28 (microlgia) PET scan
* History of fainting spells of unknown or undetermined etiology that might constitute seizures.
* History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform) EEG or immediate (1st degree relative) family history of epilepsy; with the exception of a single seizure of benign etiology (e.g. febrile seizure) in the judgment of the investigator.
* Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.).
* Metal implants (excluding dental fillings) or devices such as pacemaker, medication pump, nerve stimulator, TENS unit, ventriculo-peritoneal shunt, cochlear implant, unless cleared by the study MD.
* Substance abuse or dependence within the past six months.
* Medications will be reviewed by the responsible MD and a decision about inclusion will be made based on the following: The patient's past medical history, drug dose, history of recent medication changes or duration of treatment, and combination of CNS active drugs.
* All female participants that are pre-menopausal will be required to have a pregnancy test; any participant who is pregnant or breastfeeding will not be enrolled in the study.
* Subjects who, in the investigator's opinion, might not be suitable for the study
* A hair style or head dress that prevents electrode contact with the scalp or would interfere with the stimulation (for example: thick braids, hair weave, afro, wig)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano Santarnecchi, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Sprugnoli G, Munsch F, Cappon D, Paciorek R, Macone J, Connor A, El Fakhri G, Salvador R, Ruffini G, Donohoe K, Shafi MM, Press D, Alsop DC, Pascual Leone A, Santarnecchi E. Impact of multisession 40Hz tACS on hippocampal perfusion in patients with Alzheimer's disease. Alzheimers Res Ther. 2021 Dec 20;13(1):203. doi: 10.1186/s13195-021-00922-4. PMID 34930421

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 participants were enrolled in the study. 4 out of 5 participants completed the study. 1 study subject did not complete the follow-up amyloid and tau PET scans.
Period: Overall Study
Arm/Group | tACS
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | tACS
Number analyzed (Participants) | 5
Age, Customized [Count of Participants; unit: Participants]
  56 | 1
  64 | 1
  73 | 1
  84 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: PET Amyloid Burden
Description: Changes in the amyloid load observed via PET imaging will be evaluated by comparing PET data acquired before and after the 20 tACS sessions. The metric used is standardized uptake value ratio (SUVR), a measure of the amount of proteins in the brain identified at the PET exam. We will calculate the difference between pre and post tACS SUVR for the entire brain and report the average value (and standard deviation) for the entire group of patients. A negative value express a decrease in the amount of proteins in the brain post tACS intervention.
Time Frame: baseline and up to 12 weeks
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | tACS
Number analyzed (Participants) | 5
SUVR | -1.11 (0.76)

2. Primary Outcome: PET Tau Deposition
Description: Changes in the tau deposition observed via PET imaging will be evaluated by comparing PET data acquired before and after the 20 tACS sessions. The metric used is SUVR, a measure of the amount of proteins in the brain identified at the PET exam. We will calculate the difference between pre and post tACS SUVR (dSUVR) for the entire brain and report the average value (and standard deviation) for the entire group of patients. A negative value express a decrease in the amount of proteins in the brain post tACS intervention.
Time Frame: up to 12 weeks
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | tACS
Number analyzed (Participants) | 5
SUVR | -2.85 (1.20)

3. Secondary Outcome: PET Microglia Activation
Description: Changes in the microglia activation observed via PET imaging will be evaluated by comparing PET data acquired before and after the 20 tACS sessions. The metric used is SUVR, a measure of the amount of proteins in the brain identified at the PET exam. We will calculate the difference between pre and post tACS SUVR (dSUVR) for the entire brain and report the average value (and standard deviation) for the entire group of patients. A negative value express a decrease in the amount of proteins in the brain post tACS intervention.
Time Frame: up to 12 weeks
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | tACS
Number analyzed (Participants) | 5
SUVR | -0.56 (1.08)

4. Secondary Outcome: Changes in Brain Perfusion as Measured by Arterial Spin Labeling
Description: Patients underwent a comprehensive MRI exam before and after the tACS intervention, including measures of brain perfusion via Arterial Spin Labeling (ASL) sequences. The outcome measure represent the average change in perfusion (i.e. blood flow) recorded in regions targeted by tACS. Since Alzheimer's Disease is also characterized by a decrease of brain metabolism, an increased of blood flow after treatment would constitute a very promising sign of tACS efficacy in reducing Alzheimer's pathology in the brain.
  We will report the change in blood flow (mean, standard deviation) after tACS treatment.
Time Frame: 6 weeks (pre-post tACS intervention)
Measure: Mean (Standard Deviation); unit: mg/min/100gr
Arm/Group | tACS
Number analyzed (Participants) | 5
mg/min/100gr | 1.2 (0.6)

5. Other Pre Specified Outcome: Alzheimer's Disease Assessment Scale -Cog Score
Description: Change in Adas-Cog score will be reported, to document a potential clinical benefit of tACS. The scale ranges from 0-70 with higher score indicating greater cognitive impairment.
Time Frame: up to 12 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | tACS
Number analyzed (Participants) | 5
Scores on a scale | 1.5 (2.9)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | tACS
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tACS (N=5)
Sensation Under Electrodes (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | tACS (N=5)
Headache (General disorders) | 1
Scalp Pain (General disorders) | 2
Neck Pain (General disorders) | 1
Skin Irritation (General disorders) | 3
Sensations Under Electrodes (General disorders) | 5 — tingling, itching, burning
Visual Changes (General disorders) | 3 — flashing lights in peripheral vision
Mood Change (General disorders) | 1 — positive mood change

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT03412604/Prot_SAP_000.pdf